CLINICAL TRIAL: NCT07232914
Title: A Pilot Study of Smartphone -Based AI Assisted Ultrasound Guided Infraorbital Nerve Block in Pediatric Cleft Lip Repair : A Novel Low-cost Solution in Resource Limited Settings
Brief Title: Pilot Study of Smartphone -Based AI Assisted Ultrasound Guided Infraorbital Nerve Block in Pediatric Cleft Lip Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: O6U-ERC-0092
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Cleft Lip Repair
Keywords: AI Assisted nerve block; Cleft lip repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1:Smartphone -Based AI Assisted Ultrasound Guided Infraorbital Nerve Block (Active Comparator): Smartphone -Based AI Assisted Ultrasound Guided Infraorbital Nerve Block in pediatric cleft lip repair
  Interventions: Procedure: Infraorbital Nerve Block
- Arm 2 : Landmark based technique infraorbital nerve block (Active Comparator): Landmark based technique infraorbital nerve block in pediatric cleft lip repair
  Interventions: Procedure: Infraorbital Nerve Block

INTERVENTIONS:
Procedure: Infraorbital Nerve Block — Bilateral infraorbital nerve block smartphone based AI assisted in Arm 1 and landmark based technique in Arm 2

SUMMARY:
It's prospective single blinded randomized multi-center trial of 120 infant scheduled for primary unilateral cleft lip repair .

DETAILED DESCRIPTION:
The patients will be randomly allocated 1:1 into two groups; 60 patients in each group .AI assisted ultrasound - guided infraorbital nerve block and landmark based infraorbital nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5 -18 months
* Weight : 5-15 kilograms
* ASA I - II
* unilateral cleft lip repair

Exclusion Criteria:

* less than 5 kilograms weight
* Local infection at site of block
* Coagulopathy
* Parents refusal

Ages: 5 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Infraorbital Nerve block Success rate measured by intraoperative fentanyl consumption | Surgical incision was allowed 10 minutes after block injection
FlACC pain score | Every 6 hours postoperative for first 24 hours
  FLACC pain score (Face, Legs, Activity, Cry, and Consolability) Lower score is 0 which means no pain Highest score is 10 which means severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No